CLINICAL TRIAL: NCT00430131
Title: Investigating Best Practices for Children With Cerebral Palsy: A Pilot Study of Two Approaches
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Collaborators: Holland Bloorview Kids Rehabilitation Hospital (Other); ErinoakKids (Other)
Responsible Party: Debra Cameron, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BKR-06-055
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Last update posted 2009-08-13 (Estimated); Status verified 2009-08

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Cognitive Orientation to Occupational Performance
Procedure: Contemporary Treatment Approach

SUMMARY:
This project (CO-OP II) is the second in a series of three studies to validate a new treatment approach for children with cerebral palsy (CP). The initial study was comprised of a series of four single case studies with children with CP. It evaluated the potential of the Cognitive Orientation to Occupational Performance (CO-OP) approach to be used with children with CP and tested the procedures for CO-OP II. The overall objective of the full series of studies is to determine whether better functional outcomes are achieved for children with CP with CO-OP intervention than with contemporary occupational therapy treatment.

The primary objective of CO-OP II is to establish the feasibility of conducting a full scale randomize control trial (RCT) to discover if there are differences in functional outcomes (i.e., improvement in task performance, self efficacy) between a group of children with CP receiving CO-OP therapy and a group receiving a contemporary treatment approach (CTA). In order to meet this objective, a pilot RCT will be conducted to answer the specific research questions outlined below:

1. Do children wiht CP acquire the skills they set as goals in each of the two treatment groups?
2. Do the acquired skills generalize and transfer?
3. Are the skills maintained at 4 months post intervention?
4. Does the CO-OP approach produce a larger effect on skill acquisition and self efficacy than the CTA?
5. Does amount of parent involvement have any effect on skill acquisition or self efficacy?

Completion of this pilot RCT will provide the necessary data to conduct a full study to test the following hypothesis:

- Children with CP who receive CO-OP treatment will be more successful than children receiving CTA in improving their performance on child-chosen skills and they self efficacy.

ELIGIBILITY:
Inclusion Criteria:

* between 7 and 12 years of age
* diagnosis of cerebral palsy with hemiplegia or spastic diplegia
* Level 1,2 or 3 on the Gross Motor Function Classification Scale(GMFCS)
* normal intelligence (IQ> 85 on at least one scale (verbal or performance) of the Kaufman Brief Intelligence Test (KBIT-2)
* child assent and agreement to participate
* parental consent and agreement to participate
* sufficient language ability to communicate with and be understood during treatment

Exclusion Criteria:

* previously received or presently receiving a cognitive treatment for motor-based performance problems
* use of alternative communication system such as PECS or communication board
* regular use of BOTOX during intervention period

Ages: 7 Years to 12 Years | Sex: All
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2006-12; Study Completion 2009-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Debra L Cameron, PhD. O.T., Principal Investigator — University of Toronto